CLINICAL TRIAL: NCT04092426
Title: Prevelance of Keratoconus in Individuals Attending Refreactive Surgery Centers in Assiut
Brief Title: Prevelance of Keratoconus
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mariam hamdy, principal investigator, Assiut University
Other Study IDs: keratoconus in assiut
Record Dates: First submitted 2019-09-15; First posted 2019-09-17 (Actual); Last update posted 2019-09-17 (Actual); Status verified 2019-09

CONDITIONS: Keratoconus
MeSH Terms: conditions — Keratoconus

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- patients with keratoconus: patients with keratoconus attending refractive surgery centers in Assiut will be subjected to the following :-
  1. Full history and clinical evaluation.
  2. collection of individual data ( residency , occupation , special habbit , chronic illness )
  3. Analysis of results to assess prevelance of keratoconus and its distribution geographically in Assiut
  Interventions: Other: opthalmologic examination

INTERVENTIONS:
Other: opthalmologic examination — opthalmologic examination : Refraction Best corrected visual acuity Intraocular pressure Slit lamp examination

SUMMARY:
Keratoconus is a degenerative disease entity characterized by conical shape ectasia of the cornea. progressive conical deformation of the cornea leads to substantial astigmatism. Patients who are at an advanced stage of ectasia are often led to corneal transplant or other treatments, which essentially aim at correcting the refractive error and not in treating the ectasia. The top of the protruding cone that corneal configuration may be close to the visual axis or below and nasal of that. The disease manifests during adolescence, followed by slow progressive course, although it is possible to stabilize anytime. In 85% of cases both eyes are affected, but the severity of the attack can present significant asymmetry.

DETAILED DESCRIPTION:
Often in keratoconus a positive family history is present. Prevelance of keratoconus varies greatly worldwide.The reported prevalence of keratoconus varies widely depending upon the geographic location, diagnostic criteria used, and the cohort of patients selected. Environmental factors may contribute to the wide variation in prevalence.

the Middle East have higher prevalence than locations with cooler climates and less sunshine

ELIGIBILITY:
Inclusion Criteria:

1. persons attending refractive surgery centers in Asssiut.
2. patients found to have keratoconus are included , based on history , clinical examination and corneal topography

Exclusion criteria :

1. patients not attending those refractive surgery centers.
2. patients attending these centers but not diagnosed to be keratoconus .
3. Pregnancy or breastfeeding

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: patients with keratoconus in people attending refractive surgery
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2019-10-01 (Estimated); Primary Completion 2020-10-01 (Estimated); Study Completion 2021-10-01 (Estimated)

PRIMARY OUTCOMES:
Prevalence of keratoconus in different areas in assiut | one year
  Number of keratoconus cases detected areas in indivduals attending refractive surgery centers in Assiut

REFERENCES:
- [Background] Jonas JB, Nangia V, Matin A, Kulkarni M, Bhojwani K. Prevalence and associations of keratoconus in rural maharashtra in central India: the central India eye and medical study. Am J Ophthalmol. 2009 Nov;148(5):760-5. doi: 10.1016/j.ajo.2009.06.024. Epub 2009 Aug 11. PMID 19674732